CLINICAL TRIAL: NCT03534479
Title: Effects of Intravenous Human Polyclonal Immunoglobulins G Infusion on Endothelial Function and Insulin Sensitivity in Humans
Brief Title: Human IgGs and Endothelial Function in Vivo in Humans
Acronym: HIGH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, RAFFAELE NAPOLI, Associate Professor, Federico II University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HypoIgG1
Record Dates: First submitted 2018-05-10; First posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Common Variable Immunodeficiency
MeSH Terms: conditions — Common Variable Immunodeficiency | interventions — technetium TC 99m polyclonal IgG; Immunoglobulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CVID-IVIgG, polyclonal IgG i.v. infusion (Experimental): The patients of the CVID-IVIgG, polyclonal IgG infusion, group are studied five weeks from their last therapeutic polyclonal IgG i.v. infusion (IVIgG). On the mornings of day 0, vascular reactivity of the brachial artery, assessed as Flow mediated dilation (FMD), is measured and blood collected for biochemistry (baseline). Immediately after the FMD measurements and the blood collection, the 24 patients receive half dose of IVIgG necessary to treat their disease (400 mg/kg body weight in 10% solution). Twenty-four hours later, before infusing the second half of the dose of the IVIgG, vascular reactivity is again measured and blood collected. Vascular reactivity is again measured 1, 2, and 3 weeks after the first IVIgG infusion.
  Interventions: Drug: Polyclonal IgG

INTERVENTIONS:
Drug: Polyclonal IgG — Measurement of vascular reactivity before and after Infusion of plyclonal Immunoglobulins G in patients with Common variable immunodeficiency
  Other Names: Immunoglobulins

SUMMARY:
Endothelial dysfunction and insulin resistance play a key role in the onset and development of atherosclerosis, cardiovascular diseases, and diabetes. Data in mice models have recently demonstrated that circulating immunoglobulins G (IgG) could be involved in the process. Patients with common variable immunodeficiency (CVID), who are characterized by low circulating levels of IgG, might represent an ideal model to clarify the role played in vivo in humans by circulating IgG. Polyclonal IgG, obtained from multiple donors, given intravenously (IVIgG), are used to treat various immunodeficiencies and autoimmune diseases, including CVID. By using this disease and its treatment by IVIgG as a model, aim of the current study is to clarify whether IgG affect endothelial function and insulin sensitivity in humans in vivo and whether the action of IgG on the endothelium involves a direct interaction with the endothelial cells.

DETAILED DESCRIPTION:
For this purposes, 24 patients with CVID, receiving the last therapeutic dose of IVIgG infusion 5-weeks before the baseline measurements (CVID-IVIgG group), are studied. In all subjects, endothelial function is evaluated as flow mediated dilation (FMD) of the brachial artery, measured by ultrasonographic technique at baseline and 1, 7, 14, and 21 days after IVIgG infusion. FMD is also measured in a group of IVIgG naive CVID patients (number of patients recruited depending on availability) and a group of control healthy subjects. The latter FMD measurements serve only as a mere reference of pathological or normal values in condition of deficiency or normal levels of circulating IgG and are not used for primary outcome evaluation. To dissect further the mechanisms of improved endothelial function after IVIgG infusion, we investigate the role of human IgG on the production of Nitric Oxide (NO) in vitro on Human Coronary Artery Endothelial Cells (HCAEC) isolated from normal human coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

* Common Variable Immunodeficiency

Exclusion Criteria:

* Cancer, liver Cirrhosis, recent acute myocardial infarction, treatment with nitroderivates, Reynaud syndrome, heart failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in Endothelial Mediated Vascular Reactivity | 1 day, 1 week, 2 weeks or three weeks after polyclonal IgG infusion
  Change in vascular reactivity measured by Flow Mediated Dilation of the brachial artery

SECONDARY OUTCOMES:
Change in insulin sensitivity | 1 day, 1 week, 2 weeks or three weeks after polyclonal IgG infusion
  Change in insulin sensitivity measured as change in the Homeostasis model assessment (HOMA-IR) index

CONTACTS AND LOCATIONS:
Overall Officials: RAFFAELE NAPOLI, MD, Principal Investigator — 1990
Locations (1):
- Federico II University Hospital, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No